CLINICAL TRIAL: NCT06681584
Title: Effectiveness and Cost-effectiveness of Noninvasive Fractional Flow Reserve for Physiological Assessment in Suspected Coronary Artery Disease (ECONOMY)
Brief Title: Comparison of the Diagnostic Performance and Costs of FFRB Vs. Standard Care in Suspected Coronary Artery Disease.
Acronym: ECONOMY
Status: Active, not recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: ECONOMY; 2020/2092 (Other: SingHealth CIRB)
Record Dates: First submitted 2022-08-18; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases; Cardiovascular; Stenosis; Coronary Occlusion; Coronary Stenosis; Heart Diseases; Vascular Diseases; Constriction, Pathologic; Pathological Conditions, Anatomical
Keywords: CT angiogram; Fractional flow reserve; Coronary disease; Coronary stenosis; Coronary plaque
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Constriction, Pathologic; Coronary Occlusion; Coronary Stenosis; Heart Diseases; Vascular Diseases; Pathological Conditions, Anatomical; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA Platelet Poor Plasma , Sodium Citrate Platelet Poor Plasma and EDTA buffy coat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: Both groups of patients will receive CT scan for calcium score and Coronary angiogram, viz CTCA scan. Non-invasive FFRb will be calculated for all the patients with acceptable CTCA image quality. Based on the medical history and CTCA results, the patients may be referred for additional non-invasive tests or ICA and treated with medical therapy, PCI or CABG
  Interventions: Diagnostic Test: CTCA
- Group B: Both groups of patients will receive CT scan for calcium score and Coronary angiogram, viz CTCA scan. Non-invasive FFRb will be calculated for all the patients with acceptable CTCA image quality. However the FFRb results will only be given to the doctors who are taking care of the patients in Group B. Based on the medical history and CTCA with FFRb results (Group B), the patients may be referred for additional non-invasive tests or ICA and treated with medical therapy, PCI or CABG
  Interventions: Diagnostic Test: CTCA

INTERVENTIONS:
Diagnostic Test: CTCA — CTCA is a non-invasive test for diagnosis of anatomic coronary stenosis. Additionally, the diagnostic performance of FFRB (derived from in house calculation) with CCTA data in patients with intermediate coronary artery disease (CAD), as compared to an invasive FFR reference standard (FFR<=0.80)

SUMMARY:
Chest pain due to coronary artery disease (CAD) is a main driver of healthcare costs. Fractional flow reserve (FFR) measurement during invasive coronary angiography (ICA) is the gold standard to discriminate ischemia. A rapid simplified method had been developed to determine non-invasive FFR (FFRB) by applying computational fluid dynamics (CFD) simulation on anatomic models derived from computed tomographic coronary angiography (CTCA).In this current study, the aims is to compare the diagnostic accuracy, clinical effectiveness, safety outcomes, and quality of life of using FFRB on top of CTCA for CAD diagnosis and treatment planning, versus standard of care in Singapore; and measure health care resource utilization and assess cost-effectiveness of adopting FFRB on top of CTCA to support decision making in managing patients with suspected CAD.

DETAILED DESCRIPTION:
Chest pain due to coronary artery disease (CAD) is a main driver of healthcare costs. Fractional flow reserve (FFR) measurement during invasive coronary angiography (ICA) is the gold standard to discriminate ischemia. A rapid simplified method had been developed to determine non-invasive FFR (FFRB) by applying computational fluid dynamics (CFD) simulation on anatomic models derived from computed tomographic coronary angiography (CTCA), which compares favorably with invasive FFR and significantly improves diagnostic accuracy than CTCA alone in a previous preliminary study.

In this study, the aim is to compare the diagnostic accuracy, clinical effectiveness, safety outcomes, and quality of life of using FFRB on top of CTCA for CAD diagnosis and treatment planning, versus standard of care in Singapore; and measure health care resource utilization and assess cost-effectiveness of adopting FFRB on top of CTCA to support decision making in managing patients with suspected CAD.

The study protocol for CTCA scan is as follows.

1. CTCA will be performed with Single- or dual-source CT scanners (Toshiba AquilionOne, Cannon Aquilion One, Philips 256-dector, GE Revolution, Siemens Somatom Force Dual Source 384-detector, Siemens Somatom Drive Dual Source 256-detector) scanners.
2. CTCA scan will follow local CTCA scanning protocols that meet the quality standards defined by the Society of Cardiac Computed Tomography.
3. The CTCA image analysis will be performed according to accepted guidelines for reporting.

A total of 400 patients with chest pain will be recruited and randomly assigned into two groups. Both groups of patients will receive CTCA. But only one group of patients will be given the FFRB results. Based on the available medical information, the patients may be referred for additional non-invasive tests or ICA. For the recruited patients, who are referred for ICA subsequently, at least one FFR measurement will be conducted. All recruited patients will receive follow up at the time of 90days, 180 days and 365 days post-CTCA, as well as at the end-of-study, to record the quality of life, medical expenses and MACE events. The recruited patients will also receive follow up (phone or office visit) at the time of 90days (+30/-15 days), 180 days (+/-30 days) and 365 days (+/- 30 days) after enrolment, as well as at the end-of-study when the last recruited patient has completed one-year follow-up. Patient's response to the two questionnaires (SAQ 7 and EQ-5D-5L), their use of medication and the following clinical events will be recorded during the baseline visit and follow ups.

1. noninvasive or invasive coronary diagnostic tests;
2. planned clinic or hospital visits for evaluation or treatment of CAD;
3. unplanned hospitalization due to persisting or increasing complaints of chest pain with or without ST-T changes leading to urgent revascularization performed within the same hospitalization;
4. vascular events related to invasive diagnostic or therapeutic coronary procedures occurring within 14 days of invasive procedure;
5. nonfatal myocardial infarction;
6. Cardiovascular death defined as any death due to immediate cardiac or vascular cause or non- cardiovascular death, defined as any death not covered by the above definition. Un-witnessed death and death of unknown cause will be classified as cardiovascular death.

Through this study, investigation can be done on the clinical and cost-effectiveness of adding FFRB in the management of patients with suspected CAD. This new non-invasive method, FFRB, may help reduce the need for ICA in patients with suspected CAD and enhance the cost-effectiveness and clinical outcome of CAD diagnosis and treatment.

Once enrolled into the study, patient's medical records and medical bill/cost will also be reviewed for data collection.

For the recruited patients, who are referred for ICA subsequently (within 6 month post-CTCA) and don't have coronary revascularization or myocardial infarction event between the CTCA and ICA tests, at least one FFR measurement during ICA will be conducted.

The study protocol for ICA and FFR measurement is as follows:

1. ICA will be performed by certified interventional cardiologists following the guidelines set forth by the American College of Cardiology/ American Heart Association Task Force on Practice Guidelines and the Society for Cardiac Angiography and Interventions.
2. FFR will be performed in vessels having diameter stenosis between 30-90%, and deemed clinically indicated for evaluation.

I. Following administration of intracoronary nitroglycerin, invasive FFR will be performed using either the pressure monitoring guidewire (St Jude Medical Aeris®, Philips Volcano VerrataTM pressure wire or Boston® guidewire), or fibreoptic pressure catheter (Medtronic ACIST®) advanced distal to the stenosis.

II. Hyperemia is induced by administration of one of the following:

1. Intravenous adenosine at a rate of at least 140 mcg/kg/min; or
2. Intracoronary adenosine of at least 200 mcg into left coronary artery, and at least 100 mcg into right coronary artery;or
3. Intracoronary Papaverine of at least 20mg for the left coronary artery, and at least 15mg for the right coronary artery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 98
* Providing written informed consent
* Subjects with intermediate likelihood of obstructive CAD and with symptomatic suspected CAD who are scheduled to undergo initial clinically-indicated non-invasive coronary evaluation and have not undergone non-invasive coronary evaluation, including exercise tolerance testing, stress echocardiography, SPECT or MRI, or CTCA within the past 90 days OR ICA at any time.

Exclusion Criteria:

* Suspicion of acute coronary syndrome. Subjects experiencing unstable angina are not excluded where clinical documentation has ruled out myocardial infarctions.
* Prior, clinically documented myocardial infarction
* PCI prior to first test
* Coronary artery bypass grafting (CABG) prior to first test
* Contraindications for CTCA such as
* Presence of pacemaker or internal defibrillator leads
* Atrial Fibrillation
* Known anaphylactic allergy to iodinated contrast
* Pregnancy or unknown pregnancy status in women of childbearing potential
* Body mass index> 35kg/m2
* Contraindication to acute beta blockade

Ages: 21 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with intermediate likelihood of obstructive CAD and with symptomatic suspected CAD who are scheduled to undergo initial clinically-indicated non-invasive coronary evaluation and have not undergone non-invasive coronary evaluation, including exercise tolerance testing, stress echocardiography, SPECT or MRI, or CTCA within the past 90 days OR ICA at any time.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Compare the diagnostic performance of FFRB vs. standard care in suspected coronary artery disease. | 1 year for each enrolled subject
  The outcome is the rate of invasive coronary angiography.

SECONDARY OUTCOMES:
Compare the total costs based on FFRB compared with standard care in suspected coronary artery disease. | 1 year for each enrolled subject
  The outcome is total costs (SGD $) during 1 year follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Lohendran Baskaran, Principal Investigator — lohendran.baskaran@singhealth.com.sg
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - National Heart Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No